CLINICAL TRIAL: NCT00923494
Title: Effectiveness of Ultrasound Guided Supraclavicular Brachial Plexus Block With 20, 30, or 40 ml of Ropivacaine 0.5%
Brief Title: Effectiveness of Ultrasound (US) Guided Supraclavicular Block
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll. Change in patient population.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaime Ortiz, Assistant Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-24506
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Analgesia; Pain
Keywords: Anesthesia
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group R20 (Active Comparator): Patient will receive 20 ml of ropivacaine 0.5% for their ultrasound guided supraclavicular block.
  Interventions: Drug: 20 ml of ropivacaine 0.5%
- Group R30 (Active Comparator): Patient will receive 30 ml of ropivacaine 0.5% for their ultrasound guided supraclavicular block.
  Interventions: Drug: 30 ml of ropivacaine 0.5%
- Group R40 (Active Comparator): Patient will receive 40 ml of ropivacaine 0.5% for their ultrasound guided supraclavicular block.
  Interventions: Drug: 40 ml of ropivacaine 0.5%

INTERVENTIONS:
Drug: 20 ml of ropivacaine 0.5% — Patient will receive 20 ml of ropivacaine 0.5% for their ultrasound guided supraclavicular block.
  Arms: Group R20
Drug: 30 ml of ropivacaine 0.5% — Patient will receive 30 ml of ropivacaine 0.5% for their ultrasound guided supraclavicular block.
  Arms: Group R30
Drug: 40 ml of ropivacaine 0.5% — Patient will receive 40 ml of ropivacaine 0.5% for their ultrasound guided supraclavicular block.
  Arms: Group R40

SUMMARY:
This research study is being done in order to find out if there is any difference in the effectiveness of ultrasound guided supraclavicular brachial plexus nerve block that can be achieved with 3 different amounts of ropivacaine 0.5% (20 ml, 30 ml, and 40 ml). The investigators want to show if you can have a successful nerve block with less amount of local anesthetic, thus potentially decreasing the risk of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-64,
* Patients who are ASA I-III, presenting for distal upper extremity surgery. Surgeries to be considered are ORIF of distal upper extremity fractures such as ORIF radius, ORIF ulna, ORIF of any bones in the wrist or hand, and distal upper extremity surgery involving bones or tendons for which postoperative pain is to be expected. No emergency surgeries will be considered.

Exclusion Criteria:

* Emergency surgery,
* Patient or surgeon refusal
* Patients for which peripheral nerve block or study medications are contraindicated,
* Patients on chronic analgesic therapy at home,
* History of nerve injury, neuropathy, or known neurologic injury or illness, or inability to properly describe postoperative pain to investigators (language barrier, psychiatric disorder, dementia).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Onset of analgesia | First 30 minutes
Duration of analgesia | 24 hours

SECONDARY OUTCOMES:
Total analgesic use | First 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ortiz, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States